CLINICAL TRIAL: NCT04686474
Title: Effect of the Compound Extracted From Azadirachta Indica Leaves in the Treatment of Arsenical Keratosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Israt Zahan Zarin, MD, Resident, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BSMMU/2020/1643
Record Dates: First submitted 2020-12-23; First posted 2020-12-28 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Keratotic Nodular Size

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Azadirachta indica leaves extract containing ointment intervention. (Experimental): Azadirachta indica leaves extract containing ointment will be used twice daily for 12 weeks
  Interventions: Drug: Azadirachta indica leaves extract containing ointment intervention.

INTERVENTIONS:
Drug: Azadirachta indica leaves extract containing ointment intervention. — Azadirachta indica leaves extract containing ointment, white petroleum, bee wax, stearyl alcohol

SUMMARY:
Prepare an ointment from Azadirachta indica leaves extract and its apply on palmer arsenical keratosis patient, for 12 weeks. After intervention, effect of the ointment will be observed by measuring the nodule (before and after apply the ointment)

DETAILED DESCRIPTION:
Arsenicosis or arsenic toxicity caused by prolong ingestion of contaminated groundwater by inorganic arsenic (more than 0.05 mg/liter). It is the severest natural calamity widespread specially in Bangladesh where 61 districts out of 64 are affected. The commonest and earliest feature of arsenicosis is skin involvement like keratosis, melanosis and skin carcinoma. Keratosis of the palm and soles reduce the working ability of the patient's and affect their socio-economic condition. There is no specific treatment for keratosis. Short-term improvement may occur by using some topical keratolytic like salicylic acid, propylene glycol, eating some dietary supplementation like vitamin A, C, E, zinc, folic acid and foodstuffs like corn, spinach but symptoms recure after stoppage of these treatments. Also, these treatments require longer duration which ultimately affects patient adherence. Azadirachta indica leaves contain flavonoids, quercetin, azadirachtin, nimbin, steroids, alkaloids, phenolic compounds and other biologically active compounds that have anti-proliferative, anticarcinogenic, antioxidative and immunostimulant effects. For this reason, a study named "Effect of ethanol extract of leaves of Azadirachta indica on palmer arsenical keratosis: A single-blind trial" was done in the Department of Pharmacology, Bangabandhu Sheikh Mujib Medical University, which was found effective . So, the purpose of this study is to evaluate the effectiveness of the identified compound on moderate to severe arsenical keratosis which will be isolated from A. indica leaves extract. After IRB clearance, 35 patients with moderate to severe arsenical keratosis will be collected based on inclusion and exclusion criteria from the arsenic affected area, located at Kamalla Union of Muradnagar Upazilla, Comilla. The study will be quasi-experimental study. Included patients will be informed about the purpose of this study, as well as harmful and beneficial effects. Informed written consent, detail history, clinical examination, photographs of the palm and sole and nail samples will be collected before starting recruitment to confirm arsenicosis. For identification of isolated compounds present in the A. indica leaves, thin layer chromatography, nuclear magnetic resonance, and infrared spectrometry will be done. Cytotoxic effects of the A. indica leaves extract will be assessed by using brine shrimp bioassay. The ointment will be prepared from A. indica leaves extract and supplied to the patient at an interval of 2 weeks. Each patient will be advised to apply the ointment, with a clean fingertip by rubbing gently in the morning and night for 12 weeks. Regular monitoring will be done through phone calls and during a follow-up visit at the field level, about improvement and side effects of the ointment. Clinical improvement will be assessed by measuring the keratotic nodular size with the help of slide calipers. Statistical analysis will be done by paired t-test.

ELIGIBILITY:
Inclusion Criteria:

1. 19 to 65 years of age
2. Male and female both were included
3. Presence of palmar arsenical keratosis which nature was moderate to severe (2 to >5)
4. Used water at least more than 6 months which was contaminated with arsenic (>50 µg/L) especially for drinking purpose
5. Any drug like topical application did not received by the patient for at least last three month

Exclusion Criteria:

1. <19 and >65 years of age
2. Pregnant and breast feeding mother
3. Accept any treatment at least last three months for arsenicosis
4. Any type of skin disease like drug allergy, atopic dermatitis, psoriasis, eczema and other keratosis
5. Various systemic disease like diabetes mellitus, hepatitis, rheumatoid arthritis and others that affected the skin

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-10-20 (Actual); Primary Completion 2021-01-20 (Estimated); Study Completion 2021-02-20 (Estimated)

PRIMARY OUTCOMES:
Keratotic nodular size | 12 weeks
  Lesion size will be measured by slide calipers

CONTACTS AND LOCATIONS:
Overall Officials: Bangladesh Muradnagar Upazilla.Comilla, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Muradnagar Upazilla, Comilla, Bangladesh

IPD SHARING:
Plan to Share IPD: No